CLINICAL TRIAL: NCT06215547
Title: Medtronic Enterra II Neurostimulator
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Enterra HDE
Record Dates: First submitted 2019-09-12; First posted 2024-01-22 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-07

CONDITIONS: Gastroparesis
Keywords: nausea; vomiting
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: Medtronic - Enterra II Neurostimulator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- The Medtronic Enterra II Model 37800 Neurostimulator (Other): It is powered by a hermetically sealed hybrid cathode silver vanadium oxide (HCSVO) single-cell battery. To further protect the neurostimulator components from body fluids, the electronics and power source are hermetically sealed within an oval-shaped titanium shield. The neurostimulator case has an external insulating coating to prevent skeletal muscle stimulation at the neurostimulator implant site. An uninsulated area on one side of the neurostimulator (etched identification side) forms the indifferent electrode. The uninsulated side should be positioned away from muscle tissue. The neurostimulator has a self-sealing connector assembly with a corrosion-resistant titanium alloy body & titanium setscrews. Securing the lead system requires the use of a torque wrench which is packaged with the neurostimulator.
  Interventions: Device: Enterra HDE

INTERVENTIONS:
Device: Enterra HDE — Instructions for use Implanting physicians should have experience in the surgical and/or implantation techniques for the Enterra II system, operational and functional characteristics of the Enterra II system, 12 English 37800 2014-03 and experience in the continued management of patients by stimulation parameter adjustment. Physicians may contact Medtronic before prescribing or implanting an Enterra II system for the first time, and request a referral to a physician experienced in the use of the Enterra II system. Implanting physicians should be thoroughly familiar with all product labeling.
  Cautions:
  * When using sharp instruments near the neurostimulator, be extremely careful to avoid nicking or damaging the case, the insulation, or the connector block. Damaging the neurostimulator may require surgical replacement.
  * Do not use saline or other ionic fluids at connections, which could result in a short circuit

SUMMARY:
Humanitarian Device: Authorized by Federal (U.S.A.) Law for use in treatment of chronic intractable (drug refractory) nausea and vomiting secondary to gastroparesis of diabetic or idiopathic etiology.

DETAILED DESCRIPTION:
Description The Medtronic Enterra II Model 37800 Neurostimulator is a programmable device designed to deliver therapy through gastric electrical stimulation when connected to a lead system.

These components comprise the implantable portion of the Medtronic Enterra II system.

The operation of the neurostimulator is supported by a clinician programmer. The neurostimulator (Figure 1) operates on a sealed battery and electronic circuitry to provide controlled electrical pulse stimulation, through the implanted lead system.

A wide range of noninvasively programmable parameters and stimulation modes are available. The neurostimulator provides current parameter information, via telemetry, when used with the clinician programmer.

System Components

* Neurostimulator: Medtronic Enterra II Model 37800
* Controlling Devices: Medtronic Model 8840 Clinician Programmer with Model 8870 Application Card. Model 8527 Printer optional.
* Lead: Medtronic Enterra Model 4351 Unipolar Lead

ELIGIBILITY:
Inclusion Criteria:

* chronic intractable (drug refractory) nausea and vomiting secondary to gastroparesis of diabetic or idiopathic etiology in patients aged 18 to 70 years.

Exclusion Criteria:

* Organ transplant
* Organic obstruction
* Pseudo-obstruction
* Prior gastric surgery
* Scleroderma
* Amyloidosis
* History of seizures
* Peritoneal or unstable dialysis
* Chemical dependency
* Pregnancy
* Primary eating or swallowing disorders
* Psychogenic vomiting
* Implanted electronic medical devices
* Age < 18 or > 70 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-09-15 (Actual); Primary Completion 2025-09-14 (Estimated); Study Completion 2025-09-14 (Estimated)

PRIMARY OUTCOMES:
Treating Self Reported Nausea and Vomiting using Enterra II during procedure | Up to 30 days
  Using Enterra II system to prevent self reported Nausea and vomiting during a procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Kukreja, MD, Principal Investigator — Methodist Heath System
Locations (1):
- Methodist Richardson Medical Center, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No at this moment.